CLINICAL TRIAL: NCT05105022
Title: The Hemodynamic Effects of Propofol Versus Sevoflurane for Induction of Anesthesia in Healthy Infants as Measured by Electrical Cardiometry: Randomized Controlled Trial
Brief Title: Propofol Versus Sevoflurane for Induction of GA in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shymaa Fathy, Lecturer of anesthesia and SICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ms_203_2021
Record Dates: First submitted 2021-09-25; First posted 2021-11-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Induction of General Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Experimental): Propofol at a dose of 2mg/kg will be administered I.V. .
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): Sevoflurane (4%) will be used for inhalational induction.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous induction of general anesthesia in infants 3 months or less.

SUMMARY:
This comparative study aims to investigate the haemodynamic safety profile for induction of general anesthesia in infants 3 months or less guided by electrical cardiometry parameters versus sevoflurane.

DETAILED DESCRIPTION:
This study aims to investigate the hemodynamic effects of both propofol and sevoflurane for induction of anesthesia in infants less than 3 months of age by electrical cardiometry. The investigators hypothesized that propofol will have a safe hemodynamic profile for induction of anesthesia in infants less than 3 months of age as measured by electrical cardiometry in addition to its favorable pharmacokinetic profile of rapid induction and optimal intubation conditions.It is conducted at Abu Al Reesh Children's Hospital, Faculty of Medicine, Cairo University based on an institutional protocol used as a standard of care to induce anesthesia

ELIGIBILITY:
Inclusion Criteria:

* infants aged 3 months or less scheduled for elective surgery

Exclusion Criteria:

* significant structural congenital heart disease
* intracranial malformation.
* preexisting hemodynamic instability.
* history of seizures, opioids, and/or hypnotic administration.
* prematurity (defined as gestational age <37 weeks)

Ages: 1 Day to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
cardiac index | 15 minutes
  L/min/m2

SECONDARY OUTCOMES:
MAP | 15 minutes
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Cairo University, Cairo, Egypt